CLINICAL TRIAL: NCT03776695
Title: Phase 1 Time Lagged, Parallel-Group, Randomized, Placebo-Controlled, Single-Blind, Single Ascending Dose Study of Tyzivumab in ZIKV Infected Patients
Brief Title: Safety and Tolerability of an Antibody Against Zika Virus (Tyzivumab) in ZIKV Infected Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Zika infected patients
Sponsor: Tychan Pte Ltd. (Industry)
Collaborators: Singapore Clinical Research Institute (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ZKT-002; CTA1800062 (Other: Health Sciences Authority of Singapore)
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Treatment of Acute Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 2 mg/kg (Experimental): Subject will be administered with 2 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Biological: Tyzivumab
- 2 mg/kg - Placebo (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: Placebo
- 5 mg/kg (Experimental): Subject will be administered with 5 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Biological: Tyzivumab
- 5 mg/kg - Placebo (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: Placebo
- 10 mg/kg (Experimental): Subject will be administered with 10 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Biological: Tyzivumab
- 10 mg/kg - Placebo (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: Placebo
- 20 mg/kg (Experimental): Subject will be administered with 20 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Biological: Tyzivumab
- 20 mg/kg - Placebo (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tyzivumab — Tyzivumab Injection, (100 mg/5 mL/Vial), Zika Virus (ZIKV) Monoclonal Antibody (mAb)
  Arms: 10 mg/kg; 2 mg/kg; 20 mg/kg; 5 mg/kg
Other: Placebo — 0.9% Saline
  Arms: 10 mg/kg - Placebo; 2 mg/kg - Placebo; 20 mg/kg - Placebo; 5 mg/kg - Placebo

SUMMARY:
Zika virus (ZIKV) infection is a new emerging arbovirus disease, caused by the same vector that transmits Dengue virus, Aedes aegypti. ZIKV is a growing public health problem, rapidly spreading throughout the continents since the first epidemic was reported in the French Polynesian islands.

Currently, there are several ZIKV vaccine candidates in clinical trials. However, no ZIKV therapy (biologic or small molecule) has advanced to clinical trials. Tyzivumab will be the first therapeutic in the world, specifically targeting ZIKV, to enter clinical trials.

This is a Phase 1, time-lagged, parallel-group, randomized, placebo-controlled, single-blind, single ascending dose, Tyzivumab, ZIKV monoclonal antibody (mAb), study to be conducted in ZIKV polymerase chain reaction (PCR) positive patients.

Tyzivumab will be administered once through single IV infusion over 30 minutes. Total duration of study participation is estimated at approximately 85 days from the date of screening. Post-trial monitoring through weekly telephone calls will continue from Day 85 post-dose onwards for another three (3) more months.

The main objective of this study is to evaluate the safety of Tyzivumab in acutely infected adult patients. Assessment of time taken to achieve negative ZIKV isolation from acute ZIKV infected subjects' blood will be the study's secondary objectives.

DETAILED DESCRIPTION:
Dose escalation in this study will include 28 ZIKV-infected patients in four (4) dose cohorts.

Eligible subjects will be enrolled into dose cohorts of seven (7) subjects each. Within each dose cohort, subjects will be randomized to either Tyzivumab or Placebo Groups, with five (5) subjects receiving Tyzivumab and two (2) receiving Placebo per cohort. There will be up to four (4) dose levels / cohorts, for a total of 28 subjects. The proposed doses to be studied are 2, 5, 10, and 20 mg/kg.

Within each dose cohort, a minimum of 48-hour interval is required between Tyzivumab dosing of subject 1 and 2 and between subject 2 and 3, and a minimum of 24-hour interval is required between Tyzivumab dosing of subject 3 and 4 and between subject 4 and 5. No such time interval will be required for the Placebo dosing of subjects (i.e. a Placebo subject can be dosed concurrently with or immediately after a Tyzivumab treatment subject). Dosing of the last dose cohort (20 mg/kg) is optional if a trend of reduction in viral load and viral isolation has been observed in dose level 1 (2 mg/kg), 2 (5 mg/kg) or 3 (10 mg/kg).

Dose escalations will be guided by review of clinical signs, adverse events (AEs), and laboratory tests (including viral titre data) of the prior group (up to Day 7 after dosing) by a safety monitoring committee. Safety analysis (up to Day 7) will also be completed for the equivalent dose of ZKT-001 prior to the commencement of dosing in ZKT-002 for each specified dose.

PD, PK and ADA measurements will be conducted at various time points throughout the study. Subjects will be followed for up to approximately Day 84 safety and tolerability assessment. Serum samples for PD, PK and ADA assessments, and urine samples for PD assessments will be taken at specified time points.

ELIGIBILITY:
Inclusion Criteria:

1. Adult volunteers, aged 21 to 60, men or women

   a. Women must fulfil one (1) of the following criteria: i. Post-menopausal; either amenorrhea ≥ 12 months or follicle stimulating hormone > 40 mIU/mL ii. Surgically sterile; hysterectomy, bilateral oophorectomy, or tubal ligation iii. Women of childbearing potential participating in heterosexual sexual relations must be willing to use adequate contraception from screening day until 100 days post-infusion b. Male subjects who are non-vasectomized (or vasectomized less than six (6) months prior to dosing) and have female partners of childbearing potential must be willing to use an effective birth control method when having heterosexual intercourse, from screening day until 100 days post-infusion
2. Any one or a combination of symptoms and signs suggestive of ZIKV acute infection, presenting within 48 hours from onset
3. Positive ZIKV PCR for acute ZIKV infection
4. Subjects who are willing to comply with the requirements of the study protocol and attend scheduled visit
5. Subjects who give written informed consent approved by the Ethical Review Board governing the site
6. Satisfactory baseline medical assessment as assessed by physical examination and normal laboratory values or minor variations that are acceptable for study entry
7. Accessible vein in the forearm for blood collection

Exclusion Criteria:

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, or immunosuppressive disorders
2. Evidence of clinically significant anaemia (HB < 10 g/dL) or any other significant active haematological disease, or having donated > 450 mL of blood within the past three (3) months
3. Evidence of substance abuse, or previous substance abuse
4. Participation or planned participation in a study involving the administration of an investigational compound within the past four (4) months or during this study period
5. Planned administration of any vaccine not foreseen by the study protocol 12 weeks before first dosing day and up to four (4) months after dosing
6. Receipt of immunoglobulins and/or any blood products within nine (9) months of study enrolment or planned administration of any of these products during the study period
7. History of any reaction to monoclonal antibodies
8. Pregnant or lactating women, or women of childbearing potential who are unwilling to use adequate contraception
9. Any condition that, in the opinion of the investigator, would complicate or compromise the study or well-being of the subject

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Event (Safety and Tolerability) | 84 Days
  Presence or absence of infusion reaction (hypersensitivity / anaphylaxis / etc.) in dose cohorts.

SECONDARY OUTCOMES:
Viral Clearance Post-Tyzivumab Infusion (Efficacy) | 84 Days
  Time taken to achieve ZIKV clearance (CL) from blood via negative virus isolation in subjects acutely infected with ZIKV when given an IV infusion of Tyzivumab

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Low, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- SingHealth Investigational Medicine Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No